CLINICAL TRIAL: NCT01024179
Title: Relationship Between Initial Plaque Characteristics and Stent Surface Coverage Patterns After Sirolimus-eluting Stent Implantation Assessment by Optical Coherence Tomography
Brief Title: Relationship Between Initial Plaque Characteristics and Stent Surface Coverage Patterns
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrolling the required number of participants has made it impractical to proceed with the trial.
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Prof, Harbin Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMUOCT-PLAQUE
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
Keywords: Optical Coherence Tomography; Coronary artery disease; Chronic total occlusion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group B: CTO (Active Comparator): Chronic total occlusion
  Interventions: Device: Polymer-based sirolimus-eluting stent (Partner stent )
- Group A : Non-CTO (Active Comparator): Non-chronic total occlusion :
  1. Fibrous plaque+fibro-calcific plaque + Lipid plaque(<2 quadrants )
  2. Lipid-rich plaque ( ≥2 quadrants )
  Interventions: Device: Polymer-based sirolimus-eluting stent (Partner stent )

INTERVENTIONS:
Device: Polymer-based sirolimus-eluting stent (Partner stent ) — Partner stent (polymer-based sirolimus-eluting stent) implanted in culprit coronary artery

SUMMARY:
Vulnerable plaque characterized by thin fibrous cap and large lipid core is an independent risk factor for most of acute cardiac event. Current clinical data showed that thin-cap fibroatheroma was more frequently observed in patients with ACS than SAP. Further OCT study indicated that patients with ACS had significantly higher incidence of incomplete neointimal coverage and malapposition after DES implantation than those with SAP. These findings imply that initial native lesion characteristics may be related to different vessel response (neointimal coverage and malapposition) after stenting. However, there is little data on the relationship between plaque characteristics and vascular response to DES after stent implantation evaluated by OCT.

Therefore, this study was designed to investigate the relationship between initial plaque characteristics and stent surface coverage or late malapposition after SES implantation. The investigators will use high resolution OCT to assess the initial culprit plaque morphology and subsequent vascular response after SES stenting at the time points of post-stenting, 6 months and 12 months. IVUS will also be performed to evaluate the tissue protrusion, malapposition, vessel remodeling at the same time points.

DETAILED DESCRIPTION:
Vulnerable plaque characterized by thin fibrous cap and large lipid core is an independent risk factor for most of acute cardiac event. Current clinical data showed that thin-cap fibroatheroma was more frequently observed in patients with ACS than SAP. Further OCT study indicated that patients with ACS had significantly higher incidence of incomplete neointimal coverage and malapposition after DES implantation than those with SAP. These findings imply that initial native lesion characteristics may be related to different vessel response (neointimal coverage and malapposition) after stenting. However, there is little data on the relationship between plaque characteristics and vascular response to DES after stent implantation evaluated by OCT.

Therefore, this study was designed to investigate the relationship between initial plaque characteristics and stent surface coverage or late malapposition after SES implantation. The investigators will use high resolution OCT to assess the initial culprit plaque morphology and subsequent vascular response after SES stenting at the time points of post-stenting, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria

General Inclusion Criteria：

1. Age:18-75Y
2. Patients with stable angina or acute coronary syndrome considered suitable for coronary revascularization.
3. Patient or legal guardian understands and agrees to comply with all specified study requirements and provides written informed consent.

Angiographic Inclusion Criteria：

1. Significant coronary de novo lesion (> 70% by visual estimation).
2. Target lesion is de novo native coronary artery lesion that can be treated with 1-2 stents.
3. Reference vessel diameter of 2.5 to 4.0 mm.

Exclusion Criteria：

General Exclusion Criteria：

1. ST-segment elevation myocardial infarction within 7 days prior to the index procedure.
2. Previous CABG.
3. Life expectancy <12 months due to another medical condition.
4. Contraindication to antiplatelet therapy
5. Creatinine level more than 2.0mg/dL or ESRD.
6. Severe hepatic dysfunction (more than 3 times normal reference values).
7. Planned surgery procedure ≤ 6 months post-index procedure.
8. Known allergy to stainless steel or a history of hypersensitivity to sirolimus or structurally related compounds.
9. Female of childbearing potential with a positive pregnancy test within 7 days before the index procedure, or lactating, or intends to become pregnant during the 12 months post index procedure.
10. Patient is not clinically appropriate for OCT evaluation in the opinion of the investigator.

Angiographic Exclusion Criteria：

1. Study lesion is ostial in location (within 3.0 mm of vessel origin).
2. Study lesion involving arterial segments with highly tortuous anatomy.
3. Complex lesion morphologies (aorto-ostial, bifurcation needs two stents technique, left main, severe thrombi, heavy calcification).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To investigate the relationship between initial plaque characteristics and stent surface coverage after sirolimus-eluting stent implantation. | 6 months
  To investigate the relationship between initial plaque characteristics and stent surface coverage after sirolimus-eluting stent implantation.

SECONDARY OUTCOMES:
Relationship between tissue prolapse and initial plaque characteristics | Post-intervention
  Relationship between tissue prolapse and initial plaque characteristics
Comparison of the differences in vascular response (surface coverage and malapposition) between CTO and non- CTO lesions. | 6-month
  Comparison of the differences in vascular response (surface coverage and malapposition) between CTO and non- CTO lesions.
Late stent malapposition( by OCT and IVUS ). | 6 months
  Late stent malapposition( by OCT and IVUS ).
Relationship between initial lesion characteristics and stent surface coverage pattern after SES implantation. | 12 -month
  Relationship between initial lesion characteristics and stent surface coverage pattern after SES implantation.
Comparison of the differences in stent surface coverage between CTO and non- CTO lesions. | 12 months
  Comparison of the differences in stent surface coverage between CTO and non- CTO lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, MD.PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The second Affiliated Hospital of Harbin Medical University, Harbin, Heilong Jiang, China